CLINICAL TRIAL: NCT05170555
Title: Diagnosis of Renal Cell Carcinoma on 68Ga-PSMA PET-CT and Radioligand Therapy With 177Lu-EB-PSMA-617
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCHPSMARCC
Record Dates: First submitted 2021-12-24; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — gallium 68 PSMA-11; 177Lu-EB-PSMA-617

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA, PET/CT and 177Lu-EB- PSMA-617 therapy (Experimental): All patients diagnosed with RCC underwent 68Ga-PSMA PET/CT scan. If the PET/CT showed high PSMA expression in tumor lesions of some patients, they would intravenously injected with the dose about 1.85GBq (50 mCi) of 177Lu-EB-PSMA-617 for therapy.
  Interventions: Drug: 68Ga-PSMA; Drug: 1.85GBq (50 mCi) of 177Lu-EB-PSMA-617

INTERVENTIONS:
Drug: 68Ga-PSMA — Intravenous injection of one dosage of 74-148 MBq (2-4 mCi) 68Ga-PSMA. Tracer doses of 68Ga- PSMA will be used to image lesions of Renal Cell Carcinoma by PET/CT.
Drug: 1.85GBq (50 mCi) of 177Lu-EB-PSMA-617 — Patients were intravenous injected with the dose about 1.85GBq (50 mCi) of 177Lu-EB-PSMA-617 every 8 weeks (±1 week) for a maximum of 3 cycles.

SUMMARY:
Renal Cell Carcinoma (RCC) is the second most common tumor in urology. Considering its origination from kidney, an organ with intense physiological uptake and excretion of 68Ga-PSMA, this study aims to evaluate the uptake of 68Ga-PSMA in RCC compared to 18F-FDG in the same patients, and assess the feasibility of 177Lu-EB-PSMA-617 treatment in patients with the advanced RCC.

DETAILED DESCRIPTION:
Renal Cell Carcinoma (RCC) is the second most common tumor in urology. As one of the popular urinary tumors, the incidence rate increases by 2-4% per year. Localized RCC is generally cured by surgery, which has achieved good efficacy. However, advanced RCC are still the main factors influencing the survival of RCC patients due to its intrinsic resistance to conventional chemotherapy or radiotherapy. 18F-FDG PET/CT is considered to be a viable tool to assess RCC at initial presentation. However, FDG uptake in RCC is lower than most other solid tumors and is indistinguishable from benign lesions. So, it is necessary to find another effective way to detect RCC and its metastases. As in known, pro-angiogenic factors (VEGF, PDGF) are strongly upregulated in clear cell RCC, leading to high vascularized tumors. 68Ga-PSMA has been developed as a targeting imaging agent widely used in prostate cancer in prostate cancer. Thus, this prospective study is going to investigate whether 68Ga-PSMA PET/CT may be superior for diagnosis, therapy response assessment and follow-up of RCC than 18F-FDG PET/CT. Furthermore, peptide receptor radionuclide therapy has been widely used in the treatment of prostate cancer lesions that showed high PSMA uptake on 68Ga-PSMA PET/CT, we'll try to assess the safety and therapeutic response to 177Lu-EB-PSMA-617 in patients with RCC.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated renal cell carcinoma patients;
* 68Ga-PSMA PET/CT and 18F-FDG PET/CT within two weeks;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against PSMA
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year
  Sensitivity and Specificity of 68Ga-PSMA PET/CT for Renal Cell Carcinoma in comparison with 18F-FDG PET/CT

SECONDARY OUTCOMES:
Safety of therapy | through study completion, an average of 1 year
  the safety assessed by CTCAE v4.0

OTHER OUTCOMES:
Therapeutic effect | through study completion, an average of 1 year
  the therapeutic response assessed by PSMA PET/CT to 177Lu-EB-PSMA-617 in patients with Renal Cell Carcinoma.
Correlation between PSMA expression and SUV in PET/CT | through study completion, an average of 1 year
  to mearsure the SUVmax of RCC on PSMA PET/CT and to investigate the expression of PSMA on primary, recurrent and metastatic RCC tumour tissue using immunohistochemistry, and analyze the correlation between them.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China